CLINICAL TRIAL: NCT06199492
Title: Intelligent Optical Probe for Guiding Core Needle Biopsy Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0117; NCI-2023-11126 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Needle Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tVisio-1 (Experimental): The device collects optical coherence tomography (OCT) images in an effort to identify tumor tissue before physical samples are collected. During the biopsy, a sterilized optical imaging probe will be placed through the standard biopsy guidance needle to collect a few images of the tissue at the tip of the biopsy needle. Then the regular biopsy will continue to collect a few biopsy cores.
  Interventions: Device: tVisio-1

INTERVENTIONS:
Device: tVisio-1 — Standard of Care Biopsy

SUMMARY:
To learn if an investigational imaging device can help to identify tumor tissue before a biopsy is taken.

DETAILED DESCRIPTION:
Primary Objectives

- To determine the feasibility of using an OCT probe that will assess tumor morphology before taking a biopsy core needle. The endpoint for this objective will be the successful placement of the optical probe through the guidance needle and collection of high-quality optical coherence tomography images.

Secondary Objectives

* To assess if OCT imaging results correlate with histopathology findings.
* To assess if artificial intelligence can correctly assess tissue type based on OCT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a primary diagnosis or suspected diagnosis of malignancy and radiographic evidence of malignant lesions involving lymph node, liver or lung for which the participant was referred to IR for image-guided biopsy.
* A target lesion that meets the following criteria:
* The target lesion must be amenable to image guided biopsy
* The target lesion must be >= 1cm to ensure that the collected images will have sufficient morphological content to run the OCT image analysis Note: The collected biopsy core for the proposed study will undergo H&E staining and analysis. The AI model will determine the percentage of tumor and necrotic tissue in each image. Histology assessment will be made in the same manner to determine AI model outcome.
* Age ≥ 18 years at the time of consenting
* Life expectancy ≥ 3 months
* Platelet count >50,000/mm3 within 6 weeks of screening
* INR <1.5 within 6 weeks of screening
* If taking antiplatelet or anticoagulation medication, it must be able to be discontinued 48 hours prior to the procedure or at the discretion of the PI (e.g., aspirin, ibuprofen, LMWH preparations)
* ECOG performance status <= 2 within 6 weeks of screening.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal participants. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization.
* All lines of prior systemic therapy are permissible. Standard concurrent chemotherapy, immunotherapy, or targeted therapy are permissible.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women; women of childbearing potential unless using effective contraception as determined by the investigator.
* Absolute neutrophil count <1000 mm3 within 6 weeks of screening
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Rahul A Sheth, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org